CLINICAL TRIAL: NCT02501824
Title: Effectiveness of Anthroposophic Therapeutic Speech in Patients With Asthma in a Real-life Outpatient Setting - a Randomised, Controlled, Multicentre Cross-over Trial
Brief Title: Effectiveness of Anthroposophic Speech Therapy in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115/10
Record Dates: First submitted 2015-07-08; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- speech therapy first (Experimental): 11 sessions of speech therapy (anthroposophic therapeutic speech), then waiting phase
  Interventions: Other: anthroposophic therapeutic speech
- speech therapy second (Experimental): 10 weeks of waiting, then 11 sessions of speech therapy (anthroposophic therapeutic speech)
  Interventions: Other: anthroposophic therapeutic speech

INTERVENTIONS:
Other: anthroposophic therapeutic speech — anthroposophic therapeutic speech

SUMMARY:
Anthroposophic therapeutic speech is a complementary method that indirectly influences breathing and uses specific vowels, consonants, syllables and metres depending on the indication. The aim of this study is to test the effectiveness of anthroposophic therapeutic speech in patients with asthma regarding clinical and physiological parameters, asthma control and quality of life.

DETAILED DESCRIPTION:
Background

Breathing retraining techniques receive increased attention in the management of asthma, since the evidence for safety and usefulness of such procedures is growing. Physiotherapist-guided breathing programs, such as the Papworth method and the Buteyko method, are most systematically investigated and hence yield the best evidence of effectiveness.

Active breathing modulation techniques are frequently assigned to complementary and alternative medicine CAM, comprising of a variety of systems and modalities other than the politically dominant healthcare system.

However, patients may take a different perspective, since the prevalence of CAM use in the treatment of asthma is at a level of 20-30% among adults and 50 - 60% for children, even if rigorous estimates are being applied.

Anthroposophic therapeutic speech applies sounds and syllabic rhythm, e.g. the hexameter, for improving articulation, breathing and cardiorespiratory interaction. The method has been used for many years as a breathing retraining method for asthma in all settings. This study is the first to systematically investigate the effects of ATS in asthma patients in a real-life outpatient setting.

Objective

The following hypotheses are tested: i) anthroposophic therapeutic speech improves relevant parameters of pulmonary function in patients with asthma. ii) anthroposophic therapeutic speech reduces the use of as-needed medication in patients with asthma. iii) anthroposophic therapeutic speech improves asthma control and quality of life in patients with asthma.

Methods

The study is a randomised, controlled, multicentre, 2-period cross-over clinical trial conducted at 3 centres in Switzerland and Germany. Participants are randomly assigned in a 1:1 allocation ratio to either firstly receive 11 speech therapy sessions or to wait (control), followed by a cross-over to the other group.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 12 years
* Asthma ≥ 1 year
* Inhaling β2 agonist ≥ once weekly

Exclusion Criteria

* Not willing to perform therapy actively
* Insufficient general condition for active therapy
* COPD
* Coronary heart disease
* Oral corticosteroids
* Pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Asthma Quality of Life Questionnaire | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in spirometry | 12 weeks and 24 weeks
Asthma Control Test | Every 4 weeks until study end, expected to be 24 weeks
Peak expiratory flow in L/min | Daily until study end, expected to be 24 weeks
  Measured with peak flow meter
Days without asthma exacerbation | Daily until study end, expected to be 24 weeks
Inhaled corticosteroids in μg according to patient's diary | Daily until study end, expected to be 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wolf, Principal Investigator — Institute of Complementary Medicine, University of Bern
Locations (1):
- Institute of Complementary Medicine, University of Bern, Bern, Switzerland

REFERENCES:
- [Derived] von Bonin D, Klein SD, Wurker J, Streit E, Avianus O, Grah C, Salomon J, Wolf U. Speech-guided breathing retraining in asthma: a randomised controlled crossover trial in real-life outpatient settings. Trials. 2018 Jun 25;19(1):333. doi: 10.1186/s13063-018-2727-z. PMID 29941003